CLINICAL TRIAL: NCT06568172
Title: Randomized Phase III Trial of Neoadjuvant Immunotherapy With Response-Adapted Treatment Versus Standard-of-Care Treatment for Resectable Stage III/IV Cutaneous Squamous Cell Carcinoma (C-PRE)
Brief Title: Testing the Addition of an Immunotherapy Drug, Cemiplimab (REGN2810), Plus Surgery to the Usual Surgery Alone for Treating Advanced Skin Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCI-2024-03425; NCI-2024-03425 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-HN014 (Other: NRG Oncology); NRG-HN014 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2024-08-22; First posted 2024-08-23 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-11

CONDITIONS: Eyelid Squamous Cell Carcinoma; Recurrent Eyelid Squamous Cell Carcinoma; Recurrent Skin Acantholytic Squamous Cell Carcinoma; Recurrent Skin Clear Cell Squamous Cell Carcinoma; Recurrent Skin Lymphoepithelial Carcinoma; Recurrent Skin Spindle Cell Squamous Cell Carcinoma; Recurrent Skin Squamous Cell Carcinoma With Sarcomatoid Differentiation; Resectable Eyelid Squamous Cell Carcinoma; Resectable Skin Acantholytic Squamous Cell Carcinoma; Resectable Skin Clear Cell Squamous Cell Carcinoma; Resectable Skin Lymphoepithelial Carcinoma; Resectable Skin Spindle Cell Squamous Cell Carcinoma; Resectable Skin Squamous Cell Carcinoma With Sarcomatoid Differentiation; Skin Acantholytic Squamous Cell Carcinoma; Skin Clear Cell Squamous Cell Carcinoma; Skin Lymphoepithelial Carcinoma; Skin Spindle Cell Squamous Cell Carcinoma; Skin Squamous Cell Carcinoma With Sarcomatoid Differentiation; Stage III Head and Neck Cutaneous Squamous Cell Carcinoma AJCC v8; Stage IV Head and Neck Cutaneous Squamous Cell Carcinoma AJCC v8
MeSH Terms: interventions — Specimen Handling; cemiplimab; Radiotherapy, Image-Guided; Radiotherapy, Intensity-Modulated; Magnetic Resonance Spectroscopy; Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A central review of 40% of patients who experience a recurrence or progression that is considered a primary endpoint event will be conducted once the number of events for the primary endpoint has been reached. Each case will be reviewed by two independent reviewers who are blinded to the patient's assigned treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (surgery, radiation) (Active Comparator): Patients undergo surgery per standard of care within 6 weeks of randomization. Starting within 6-12 weeks of surgery, patients may undergo IGRT with IMRT for 5 fractions per week for 6 weeks as clinically indicated. Patients also undergo CT, MRI, and/or PET/CT prior to treatment, and CT and/or MRI during follow up. Patients may also undergo optional collection of tissue, whole blood, and plasma on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Radiation: Image Guided Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Procedure: Surgical Procedure
- Arm 2 (cemiplimab, surgery, radiation) (Experimental): Patients receive cemiplimab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo response-adaptive surgery 21 days after last dose of cemiplimab. Starting within 12 weeks of surgery, patients may undergo IGRT with IMRT for 5 fractions per week for 6 weeks as clinically indicated. Starting within 6 weeks of completion of surgery or radiation therapy (if indicated), patients without pCR receive cemiplimab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 42 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, MRI, and/or PET/CT prior to treatment, and CT and/or MRI on study and during follow up. Patients may also undergo optional collection of tissue, whole blood, and plasma on study.
  Interventions: Procedure: Biospecimen Collection; Biological: Cemiplimab; Procedure: Computed Tomography; Radiation: Image Guided Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Procedure: Surgical Procedure

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood and/or plasma
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: Cemiplimab — Given IV
  Other Names: Cemiplimab RWLC; Cemiplimab-rwlc; Libtayo; REGN 2810; REGN-2810; REGN2810
  Arms: Arm 2 (cemiplimab, surgery, radiation)
Procedure: Computed Tomography — Undergo CT and/or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Radiation: Image Guided Radiation Therapy — Undergo IGRT
  Other Names: IGRT; Image Guided Radiotherapy; image-guided radiation therapy; Image-Guided Radiotherapy
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity modulated radiation therapy (procedure); Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Other: Questionnaire Administration — Ancillary studies
Procedure: Surgical Procedure — Undergo surgery per SOC
  Other Names: Operation; Surgery; Surgery Type; Surgery, NOS; Surgical; Surgical Intervention; Surgical Interventions; Surgical Procedures; Type of Surgery
  Arms: Arm 1 (surgery, radiation)
Procedure: Surgical Procedure — Undergo response-adaptive surgery
  Other Names: Operation; Surgery; Surgery Type; Surgery, NOS; Surgical; Surgical Intervention; Surgical Interventions; Surgical Procedures; Type of Surgery
  Arms: Arm 2 (cemiplimab, surgery, radiation)

SUMMARY:
This phase III trial compares the effect of adding cemiplimab to standard therapy (surgery with or without radiation) versus standard therapy alone in treating patients with stage III/IV squamous cell skin cancer that is able to be removed by surgery (resectable) and that may have come back after a period of improvement (recurrent). The usual treatment for patients with resectable squamous cell skin cancer is the removal of the cancerous tissue (surgery) with or without radiation, which uses high energy x-rays, particles, or radioactive seeds to kill cancer cells and shrink tumors. Immunotherapy with monoclonal antibodies, such as cemiplimab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Cemiplimab has been approved for the treatment of skin cancer that has spread or that cannot be removed by surgery, but it has not been approved for the treatment of skin cancer than can be removed by surgery. Adding cemiplimab to the usual treatment of surgery with or without radiation may be more effective in treating patients with stage III/IV resectable squamous cell skin cancer than the usual treatment alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if neoadjuvant immunotherapy combined with response-adapted oncologic surgery improves site-reported event-free survival (EFS) compared to standard-of-care surgery in resectable stage III/IV cutaneous squamous cell carcinoma (CSCC).

SECONDARY OBJECTIVES:

I. To compare utilization of adjuvant radiation between arms. II. To compare disease-free survival (DFS) between arms. III. To compare overall survival (OS) between arms. IV. To compare adverse events (Common Terminology Criteria for Adverse Events [CTCAE] version [v]5.0) between arms.

V. To assess pathologic complete response in arm 2.

PATIENT-REPORTED OUTCOMES:

I. Compare changes in patient reported quality of life as measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) at 1, 6, and 12 months after surgery between treatment arms. (Primary objective) II. To compare patient reported symptoms functioning, and quality of life, as measured by the Cutaneous Squamous Cell Carcinoma NeoAdjuvant, Adjuvant and Perioperative 32 question scale (CSCC NAAP-32), Patient Reported Outcomes Measurement Information System (PROMIS)-Short Form (SF)-Anxiety, PROMIS-SF-Fatigue, and EuroQol-5D (EQ-5D), between arms at 1, 6, and 12 months after surgery.

III. Develop a scoring algorithm and validate the CSCC-NAAP-32 for use in this patient population.

EXPLORATORY OBJECTIVES:

I. To compare disease-specific survival (DSS) between arms. II. To correlate pathologic response with DFS in arm 2. III. To assess overall response rate (ORR) in arm 2. IV. To compare patterns of failure between arms. V. To compare pathologic measurements of lymph node yield between arms. VI. To compare primary tumor specimen dimensions and volume between arms.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM 1: Patients undergo surgery per standard of care within 6 weeks of randomization. Starting within 6-12 weeks of surgery, patients may undergo image-guided radiation therapy (IGRT) with intensity modulated radiation therapy (IMRT) for 5 fractions per week for 6 weeks as clinically indicated. Patients also undergo computed tomography (CT), magnetic resonance imaging (MRI), and/or positron emission tomography (PET)/CT prior to treatment, and CT and/or MRI during follow up. Patients may also undergo optional collection of tissue, whole blood, and plasma on study.

ARM 2: Patients receive cemiplimab intravenously (IV) over 30 minutes on day 1 of each cycle. Cycles repeat every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo response-adaptive surgery 21 days after last dose of cemiplimab. Starting within 12 weeks of surgery, patients may undergo IGRT with IMRT for 5 fractions per week for 6 weeks as clinically indicated. Starting within 6 weeks of completion of surgery or radiation therapy (if indicated), patients without pathologic complete response (pCR) receive cemiplimab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 42 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, MRI, and/or PET/CT prior to treatment, and CT and/or MRI on study and during follow up. Patients may also undergo optional collection of tissue, whole blood, and plasma on study.

After completion of study treatment, patients are followed up at 1, 6, and 12 months post-surgery then every 3 months for 2 years, every 6 months in year 3, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of invasive cutaneous squamous cell carcinoma (CSCC) or regional lymph node or in-transit metastasis of CSCC

  * The following CSCC subtypes are eligible according to World Health Organization (WHO) classification if the predominant histology is confirmed CSCC.

    * Spindle cell squamous cell carcinoma (SCC)
    * Squamous cell carcinoma with sarcomatoid differentiation
    * Acantholytic SCC
    * Clear cell SCC
    * Lymphoepithelial carcinoma

      * Note: Keratoacanthoma SCC and Verrucous SCC subtypes are not eligible.
  * For patients with regional metastasis without a primary tumor at screening: a clinical history of CSCC that drains to the involved regional lymph nodes or in-transit metastases in question is required

    * For example, a parotid mass shown to be SCC by cytologic analysis of a fine needle aspirate in a patient with a clinical history of CSCC on the ipsilateral scalp would be eligible
  * For patients with regional metastases without a primary tumor and an ambiguous clinical history: tumor genomic sequencing suggesting a primary tumor of cutaneous origin would be acceptable evidence to establish eligibility
  * NOTE: Tumor genomic sequencing is not required to determine eligibility, but may be part of the routine evaluation of patients with cancers of unknown primary at some institutions. For example, a parotid mass shown to be SCC by cytologic analysis of fine needle aspirate without a primary tumor and an ambiguous clinical history, but with a tumor genomic sequencing assay demonstrating a high tumor mutation burden (≥ 10 mutations/Mb) and/or a high fraction of ultraviolet (UV) related mutations (> 50% of mutations [cytosine (C)/thymine (T)]C > T or CC > TT) and/or the presence of "signature 7" mutations would be eligible (Chang 2021)
* Previously untreated or recurrent CSCC
* Clinical American Joint Committee on Cancer (AJCC) 8th Edition (eyelid, head and neck sites) or Union for International Cancer Control (UICC) (non-head and neck sites) stage III or IV
* Primary tumor site must be in the head and neck cutaneous region, other non-head and neck cutaneous regions, or eyelid cutaneous region
* No mucosal squamous cell carcinoma (vermillion lip, nasal, oral, sinonasal, conjunctival, anogenital)
* Tumor must be resectable with curative intent. Note: Tumor with bony skull base invasion and/or skull base foramen involvement (T4b) is not eligible. (Patients with T4b eyelid tumors using UICC Staging, and not involving the brain, are eligible.)
* At least 1 lesion that is measurable by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* No definitive clinical or radiologic evidence of distant metastatic disease (M1), visceral and/or distant nodal disease
* Age ≥ 18
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Not pregnant and not nursing

  * Negative urine or serum pregnancy test (in persons of childbearing potential) within 14 days prior to registration. Childbearing potential is defined as any person who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal
* Absolute neutrophil count (ANC) ≥ 1,000 cells/mm^3
* Platelets ≥ 75,000 cells/mm^3
* Hemoglobin ≥ 8.0 g/dl (Note: The use of transfusion or other intervention to achieve hemoglobin [Hgb] ≥ 8.0 g/dl is acceptable)
* Creatinine clearance (CrCL) > 30mL/min by the Cockcroft-Gault formula
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (NOTE: For patients with Gilbert's syndrome, total bilirubin ≤ 3 x ULN. Gilbert's syndrome must be documented appropriately as past medical history.)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≤ 3 x institutional ULN
* No prior systemic therapy for the study cancer (including patients currently receiving immunotherapy for a separate malignancy)
* No prior radiotherapy to the region of the study cancer that would result in cumulative doses of radiation to organs at risk for radiation injury that exceed protocol limitations
* No history of myocardial infarction/unstable angina within the last 6 months
* New York Heart Association functional classification IIb or better (New York Heart Association [NYHA] functional classification III/IV are not eligible) (Note: Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association functional classification)
* No active infection requiring systemic antibiotics, antiviral, or antifungal treatments
* No history of allogeneic stem cell transplantation, or autologous stem cell transplantation
* No history of a solid organ transplant (other than corneal transplant)
* No active, known, or suspected autoimmune disease

  * Active or known disease is defined as:

    * Requiring higher than physiologic steroid levels (> 10mg prednisone/day or equivalent) or
    * Requiring disease-modifying agents or
    * Ongoing or recent (within 5 years prior to registration) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments, which may suggest risk for immune-related adverse events (irAEs)
  * NOTES:

    * Patients meeting the following criteria are not considered immunosuppressed and are eligible to enroll:

      * Patients who require a brief course of steroids (eg, prophylaxis for imaging assessments due to hypersensitivity to contrast agents) are not excluded
      * Patients with type I diabetes mellitus, and endocrinopathies (including hypothyroidism due to autoimmune thyroiditis) only requiring hormone replacement, or skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
      * Physiologic replacement doses ≤ 10 mg prednisone/day or equivalent allowed, as long as they are not being administered for immunosuppressive intent. Inhaled or topical steroids are permitted
    * Patients with the following immunosuppressed conditions are eligible to enroll:

      * Patients with HIV infection on effective anti-retroviral therapy with undetectable viral load within 6 months prior to registration are eligible
      * Patients with chronic lymphocytic leukemia (CLL) with no history of anti-CLL therapy within 6 months prior to registration are eligible
* No history of interstitial lung disease (eg, idiopathic pulmonary fibrosis, organizing pneumonia)
* No active, noninfectious pneumonitis requiring immune-suppressive therapy
* No active tuberculosis
* No live vaccines within 28 days prior to registration
* No history of allergic reaction to the study agent, compounds of similar chemical or biologic composition to the study agent (or any of its excipients)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2031-08-14 (Estimated); Study Completion 2031-08-14 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | Up to 6 years
  Defined as the time from randomization to any of the following events: progression of disease that precludes surgery, toxic effects related to treatment that preclude surgery, inability to resect all gross disease), disease recurrence (local, regional, or distant) after surgery (or after radiographic complete response), disease progression after radiographic partial response or stable disease without surgery (or biopsy, as applicable), or death due to any cause, whichever occurs first. EFS rates will be estimated using the Kaplan-Meier method, and the stratified log-rank test will be used to assess whether perioperative immunotherapy (neoadjuvant/adjuvant) with response-adapted oncologic surgery improves EFS as recorded by the site compared to standard-of-care surgery in resectable stage III/IV cutaneous squamous cell carcinoma (CSCC).

SECONDARY OUTCOMES:
Utilization of adjuvant radiation | Up to 6 years
  Rates of utilization of adjuvant radiation for each arm will be computed using a binomial distribution assumption. A 95% confidence interval (CI) for the rate difference between arms will be calculated using the stratified Newcombe (Wilson) method (Yan 2010).
Disease-free survival (DFS) | From randomization to recurrent or death, assessed up to 6 years
  DFS will use the same analytic methods as EFS.
Overall survival (OS) | From randomization to death, assessed up to 6 years
  OS will use the same analytic methods as EFS.
Incidence of adverse events | At 30 days and then up to 6 years
  Adverse events (AEs) will be graded using Common Terminology Criteria for Adverse Events version (v) 5.0. Counts and frequencies of all AEs by grade will be provided by each treatment arm. For the experimental arm, AEs will be summarized for each treatment phase (neoadjuvant, adjuvant, and post-treatment [after adjuvant]). Counts and frequencies will be provided for the worst grade AE experienced by the patient by treatment arm. The proportion of patients with at least one grade 3 or higher AE, serious AEs, AEs leading to discontinuation or death will be reported for each treatment arm. These analyses will be descriptive.
Pathologic complete response | At 1 and 2 years
  Site-reported pathologic response will be assessed using the following categories: pathological complete, major, and partial response, no pathological response (i.e., no complete, major, or partial response), and no pathological evaluation. Pathological responses at 1 and 2 years will be summarized using frequencies and percentages and tested using a chi-square test at a two-sided 5% significance level.

OTHER OUTCOMES:
Quality of life | From baseline up to 12 months after surgery
  The primary patient-reported outcome (PRO) is the global health status score as measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30. For all PRO scheduled assessment visits, patient disposition will be summarized. PRO completion rate and available data rate will be computed and reported at each timepoint. Mixed effects model with repeated measures (MMRM) will be performed for the global health status score incorporating all PRO assessment timepoints. The adjusted means for each treatment and the estimated treatment differences for the treatment comparisons will be presented together with 95% CIs.
Validation and scoring of Cutaneous Squamous Cell Carcinoma NeoAdjuvant, Adjuvant and Perioperative 32 question scale (CSCC NAAP-32) | From baseline up to 12 months after surgery
  Item response distributions, inter-item correlations, factor analysis and internal consistency will be assessed. Confirmatory factor analyses will be used to confirm the underlying structure hypothesized by the conceptual framework. Items capturing perceptions and effect of treatments will be evaluated with single-item scores. Completion rate and available data rate will be computed and reported at each timepoint. CSCC-NAAP-32 item responses will be described at baseline to evaluate floor/ceiling effects, missingness, outliers, and multi-modal distributions. Internal consistency reliability for multi-item scales will be evaluated at baseline using both Cronbach's alpha and McDonald Omega coefficients. Test-retest reliability will be assessed using intraclass correlation coefficients between two time points. Construct validity and ability to detect change over time will be assessed.
Change in patient-reported symptoms, functioning, and quality of life | From baseline up to 12 months after surgery
  PRO instruments will be scored based on their respective scoring algorithms. Descriptive statistics, MMRMs, and assessment of missing data will be performed.
Disease-specific survival (DSS) | From randomization to death due to study cancer, date of precluding event, or last follow up, assessed up to 6 years
  The cause-specific log-rank test and cause-specific Cox models will also be used to compare cause-specific HRs between treatment arms and estimate cause-specific treatment-effect HRs, respectively. The cumulative incidence method will be used to estimate the incidence of cancer-specific mortality with between-arm differences tested using the stratified Gray's test. Stratified sub-distribution HR and 95% CI for treatment effect from Fine-Gray models will be computed to supplement the DSS analysis.
Pathologic response | Up to 6 years
  Will evaluate the association of pathologic response with DFS in the experimental arm. Will compare EFS between patients with complete response versus others (major/partial/no response/not evaluable) using a log-rank test. DFS rates for each pathological response subgroup will be estimated using the Kaplan-Meier method. Furthermore, DFS rates for each pathological response subgroup will be calculated using the Kaplan-Meier method as an exploratory analysis.
Overall response rate | Up to 6 years
  Will be assessed using Response Evaluation Criteria in Solid Tumors v. 1.1 and summarized by time-point using frequencies and relative frequencies. The best objective response (complete response + partial response) rate will be estimated using a 95% confidence interval obtained using the normal approximation for a binomial proportion.
Failure patterns | Up to 6 years
  Failure patterns (local, regional, and distant metastasis) for EFS will be summarized for each treatment arm.
Lymph node yield | At time of surgery
  The pathologic measurements of lymph node yield (i.e., number of lymph nodes) will be compared between arms using the Mann-Whitney test.
Primary tumor specimen dimensions | At time of surgery
  The pathologic measurements of the primary tumor specimens' length, width, and volume will be compared between arms using the t-test for independent samples. A Mann-Whitney test will be used if the distribution of a variable does not pass the normality test.
Treatment effect HR estimates | Up to 6 years
  Treatment effect HR estimates and 95% CIs for the primary and secondary endpoints (EFS, DFS, DSS, OS) will be calculated using a (cause-specific) Cox model with treatment by factor interaction for the following subgroups:
  * Immunosuppressed (Yes versus [vs.] no)
  * Advanced nodal disease (N3 or in-transit metastases vs. other).
  * Clinical Union for International Cancer Control or American Joint Committee on Cancer 8th Edition stage III vs. IV
  * Female vs. male
  * Age < 70 vs. ≥ 70 years
  * Eastern Cooperative Oncology Group performance status (0 vs. 1-2)
  * Females vs. males
  * White vs. other race
  * Head and neck vs. trunk/extremities
  * T stage (Tx-2 vs. > T2)
  * N stage (N0-1 vs. > N1)
  * Country A forest plot with these treatment effect HR estimates will be provided.
Treatment effect estimates by sex | Up to 6 years
  Estimates of the primary outcome treatment effect and the corresponding 95% CIs by sex will be provided.
Treatment effect estimates by race | Up to 6 years
  Estimates of the primary outcome treatment effect and the corresponding 95% CIs by race will be provided.
Treatment effect estimates by ethnicity | Up to 6 years
  Estimates of the primary outcome treatment effect and the corresponding 95% CIs by ethnicity will be provided.

CONTACTS AND LOCATIONS:
Overall Officials: Neil D Gross, Principal Investigator — NRG Oncology
Locations (187):
- United States (182):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Tower Cancer Research Foundation, Beverly Hills, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UC San Diego Health System - Encinitas, Encinitas, California
  - City of Hope at Irvine Lennar, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - City of Hope Antelope Valley, Lancaster, California
  - The Angeles Clinic and Research Institute - West Los Angeles Office, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - City of Hope South Pasadena, South Pasadena, California
  - Torrance Memorial Physician Network - Cancer Care, Torrance, California
  - City of Hope Upland, Upland, California
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Yale University, New Haven, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - UM Sylvester Comprehensive Cancer Center at Doral, Doral, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - Sarasota Memorial Hospital-Venice, N. Venice, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Florida Cancer Specialists - Sarasota, Sarasota, Florida
  - Florida Cancer Specialists - Sarasota Downtown, Sarasota, Florida
  - First Physicians Group - Silverstein Institute at Floyd Street, Sarasota, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Sarasota Memorial Health Care Center at University Parkway, Sarasota, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Florida Cancer Specialists - Venice Pinebrook, Venice, Florida
  - Florida Cancer Specialists - Venice Island, Venice, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Alton Memorial Hospital, Alton, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - IU Health North Hospital, Carmel, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Heartland Oncology and Hematology LLP, Council Bluffs, Iowa
  - Methodist Jennie Edmundson Hospital, Council Bluffs, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - University of Michigan - Brighton Center for Specialty Care, Brighton, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MECC, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - SUNY Upstate Medical Center-Community Campus, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - Atrium Health Stanly/LCI-Albemarle, Albemarle, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - Atrium Health University City/LCI-University, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Levine Cancer Institute-Gaston, Gastonia, North Carolina
  - Atrium Health Union/LCI-Union, Monroe, North Carolina
  - Duke Cancer Center Raleigh, Raleigh, North Carolina
  - Atrium Health Cleveland/LCI-Cleveland, Shelby, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - UH Seidman Cancer Center at UH Avon Health Center, Avon, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - Saint Vincent Hospital, Erie, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Rock Hill Radiation Therapy Center, Rock Hill, South Carolina
  - Levine Cancer Institute-Rock Hill, Rock Hill, South Carolina
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - MD Anderson in The Woodlands, Conroe, Texas
  - UT Southwestern Simmons Cancer Center - RedBird, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - William S Middleton VA Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Drexel Town Square Health Center, Oak Creek, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
- Australia (3):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- Canada (2):
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm